CLINICAL TRIAL: NCT03098368
Title: Rotigotine Effect on Nocturnal Hypokinesia Compares to Placebo Control: A Quantitative Assessment by Wearable Sensors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JSringean
Record Dates: First submitted 2017-02-13; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Nocturnal Hypokinesia
Keywords: Parkinson's disease; Rotigotine transdermal patch; Nocturnal hypokinesia
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine; Control Groups

STUDY DESIGN:
Intervention Model Description: Active group is the group of PD patients who received rotigotine transdermal patch titration from 2 mg/day to maximum effect dose which participants had no side effect or reach 16 mg/day every week.
  Placebo group is the group of PD patients who received the placebo patch titration every week the same protocol as the active group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The active drugs and placebo were labeled from the company and the study nurse would give the drug to participants who were randomized.

ARMS (2):
- Patient (active) group (Active Comparator): * Rotigotine titration up to 16 mg/24 hr
  * Starting dose 2 mg/24 hr up titrate 2 mg weekly to optimal/maximum dose
  * Duration up to 12 weeks
  * The treatment was titrated until optimal dosage
    * (that which patient/ caregiver felt that nocturnal hypokinesia and/or early morning akinesia was adequately controlled)
    * (or patient can not tolerated the side effects such as dyskinesia)
  * All previous dopaminergic medications were not allowed to adjusted during the study period.
  Interventions: Drug: Rotigotine
- Control (placebo) group (Placebo Comparator): Placebo transdermal patch were titration with the same protocol as active group.
  Duration up to 12 weeks
  * The treatment (placebo patch) was titrated until optimal dosage
    * (that which patient/ caregiver felt that nocturnal hypokinesia and/or early morning akinesia was adequately controlled)
    * (or patient can not tolerated the side effects such as dyskinesia)
  * All previous dopaminergic medications were not allowed to adjusted during the study period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotigotine
  Other Names: Neupro patch
  Arms: Patient (active) group
Drug: Placebo — Placebo of rotigotine patch
  Other Names: Control group
  Arms: Control (placebo) group

SUMMARY:
Parkinson's disease (PD) is the neurodegenerative disease which is caused by Lewy bodies deposition in central and peripheral nervous system. The mains symptoms include both motor and non motor symptoms such as bradykinesia, rigidity, rest tremor, postural instability, autonomic dysfunction or neuropsychiatric symptoms. Moreover, the PD symptoms not only occur in the daytime, but also in the nighttime. The nighttime symptoms or nocturnal symptoms can make the patients disabling as well as the daytime symptoms. The bradykinesia that occurs in the nighttime is called nocturnal hypokinesia which also make many serious consequences such as bedsore, falling or aspiration or death.

In this study, the investigators aim to study the effects of rotigotine transdermal patch compare to placebo on mainly the aspect of nocturnal hypokinesia.

DETAILED DESCRIPTION:
The investigators recruited PD patients who had history of nocturnal hypokinesia and randomized by running number (blind) into 2 groups including active and placebo group. Baseline demographic, disease characteristics, nocturnal questionnaires and wearable nocturnal sensors data were collected before drug titration. In active group, participants received the rotigotine transdermal patch titration from 2 mg/day to maximum dosage which participants had no side effect or 16 mg/ day every week. In placebo group, participants would get the placebo patch titration as the active group. After participants got maintenance dosage, participants would get the physical examination, nocturnal questionnaires and wearable nocturnal sensors as before study.

ELIGIBILITY:
Inclusion Criteria:

* Patients: PD patients (age ≥ 18 years) who have history of nocturnal hypokinesia
* Patients not taking levodopa were eligible for study
* Patients who taking immediate- released levodopa,they had been on a stable dose for 28 days prior to baseline assessment and during the study
* Patients did not use control-released L-dopa at bedtime

Exclusion Criteria:

* History of narcolepsy, excessive daytime sleepiness, sudden onset of sleep
* History of hallucination, dementia and psychosis
* Evidence of ICDs
* Clinical relevant to cardiovascular disorders (including prolonged QTc ≥ 500 ms, recent MI)
* History of seizure or stroke in the past 1 year
* Patients had participated in other clinical trial in the past 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Nocturnal parameters from wearable sensors during nighttime | up to 10 hours
  The wearable sensors are the tri-axis accelerometer and gyrometer which will be attached at waist and wrist of patients up to 10 hours. The raw data from wearable sensors will be analyzed by MATLAB program. The results from MATLAB include the number of turning in bed.

SECONDARY OUTCOMES:
Nocturnal Akinesia Dystonia Cramp score (NADCs) | Before and after maintenance dosage intervention within 1 month.
  The nocturnal akinesia dystonia cramp score (NADCs) questionnaire was asked before and after participants got the interventions in both active and placebo groups.
PDSS-2 | Before and after maintenance dosage intervention within 1 month.
  The Parkinson's disease sleep scale- 2 questionnaire was asked before and after participants got the interventions in both active and placebo groups.